CLINICAL TRIAL: NCT00986349
Title: A Phase II Single-Center, Prospective, Open Label Efficacy Study, of the GI EndoBarrier™ Liner for the Treatment of Type 2 Diabetes
Brief Title: Study of EndoBarrier Liner for Treatment of Type 2 Diabetes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Morphic Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-2
Record Dates: First submitted 2009-09-27; First posted 2009-09-29 (Estimated); Results first posted 2017-01-02 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-01

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Weight Loss; GI Dynamics; EndoBarrier
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diabetes (Experimental): Single Arm
  Interventions: Device: EndoBarrier Liner

INTERVENTIONS:
Device: EndoBarrier Liner — 52 week treatment of EnoBarrier Liner
  Other Names: EndoBarrier Gastrointestial Liner; GI Sleeve

SUMMARY:
The main objective of the study is to demonstrate the safety and efficacy of the Gastrointestinal (GI) EndoBarrier in the glycemic control of diabetes in subjects with Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects Age > 18 years and ≤ 55 years
* Male or Female
* Subjects with Type 2 Diabetes who have been treated for ≤10 years and are on oral diabetic medications
* Subjects with an HbA1C > 7.5 and ≤ 10.0%
* Subjects with a BMI > 26 - < 50
* Subjects willing to comply with study requirements
* Subjects who have signed an informed consent form
* Women who are post-menopausal, surgically sterile or on oral contraceptives and agree to remain on oral contraceptives for at least twenty-four (24) weeks after being implanted or the duration of their trial participation and agree not to become pregnant during the trial.

Exclusion Criteria:

* Subjects diagnosed with Type 1 Diabetes Mellitus or having a history of ketoacidosis
* Subjects requiring insulin
* Subjects with probable insulin production failure (fasting C Peptide serum <1ng/mL)
* Subjects that have autoimmune disease as evidenced by a positive anti-GAD blood test
* Subjects with a weight loss of > 4.5 Kg (10 lbs) within the 12 Weeks of screening
* Subjects requiring prescription anticoagulation therapy
* Subjects with or a history of iron deficiency and/or iron deficiency anemia
* Subjects with or a history of abnormalities of the GI tract
* Subjects with symptomatic gallstones or kidney stones at the time of screening
* Subjects with a known infection
* Subjects with or a history of coagulopathy, upper gastro-intestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasia
* Subjects mentally retarded or emotionally unstable, or exhibits psychological characteristics which, in the opinion of the Investigator, makes the Subject a poor candidate for device placement or clinical trial participation
* Subjects with previous GI surgery that could affect the ability to place the device or the function of the implant
* Subjects unable to discontinue NSAIDs (non-steroidal anti-inflammatory drugs) during the implant period
* Subjects with active H. pylori (Note: Subjects may be enrolled if they had a prior history of H. Pylori and were successfully treated)
* Subjects receiving weight loss medications such as Meridia, Xenical, or over the counter weight loss medications
* Subject or Family history of a known diagnosis or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder
* Subjects with active and uncontrolled GERD
* Subjects with a known history of substance abuse
* Subjects participating in another ongoing investigational clinical trial
* Subjects taking corticosteroids or drugs known to affect GI motility (i.e. Reglan)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Cohen, MD, Principal Investigator — Hospital Alemão Oswaldo Cruz
Locations (1):
- Hospital Alemão Oswaldo Cruz, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data is on file at the Sponsor

RESULTS

PARTICIPANT FLOW:
Groups:
- EndoBarrier Liner Device: Enrolled Subjects
Period: Overall Study
Arm/Group | EndoBarrier Liner Device
Started | 23 (attempted implant procedures)
Successful Implant Procedure (Three subjects had anatomy that could not accommodate the device implant) | 20 (successful device implant procedure)
Early Explant | 4
Completed | 16
Not Completed | 7
Not completed — Unsuccessful implant procedure | 3
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1
Not completed — device migration | 1

BASELINE CHARACTERISTICS:
Population: Subjects with successful implants
Groups:
- EndoBarrier Liner Device: EndoBarrier Liner: 52 week treatment of EndoBarrier Liner
Arm/Group | EndoBarrier Liner Device
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (6.69)
Gender [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Region of Enrollment [Number; unit: participants]
  Brazil | 20

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Glycemic Control (HbA1c) Over Time
Description: HbA1c (%) at Baseline, Month 3, Month 6, Month 9, and Month 12
Time Frame: Baseline to 12 Months with device implanted
Population: 20 subjects with a successfully implanted device were analyzed at Baseline. 1 subject removed at day 75 due to non-compliance with attending required visits. 1 subject removed at 175 due to device rotation, 2 subjects removed at day 203 and 313 due to abdominal pain AE
Measure: Median (Full Range); unit: HbA1c %
Groups:
- EndoBarrier Liner Device at Baseline: HbA1c %
- EndoBarrier Liner Device at 3 Months: HbA1c % One subject was removed at day 75 due to non-compliance with attending required visits.
- EndoBarrier Liner Device % at 6 Months; EndoBarrier Liner Device % at 9 Months; EndoBarrier Liner Device % at 52 Weeks: HbA1c
Arm/Group | EndoBarrier Liner Device at Baseline | EndoBarrier Liner Device at 3 Months | EndoBarrier Liner Device % at 6 Months | EndoBarrier Liner Device % at 9 Months | EndoBarrier Liner Device % at 52 Weeks
Number analyzed (Participants) | 20 | 19 | 19 | 17 | 16
HbA1c % | 8.7 [7.4 to 10.2] | 6.7 [5.7 to 9.4] | 6.9 [5.8 to 8.9] | 6.9 [5.9 to 9.3] | 6.8 [5.9 to 11.0]

2. Primary Outcome: Change in Anti-diabetes Medications
Description: Medications were classified as "increased" if the dose of one or more oral agents was higher or an additional glucose-lowering agent was utilized at the time of treatment completion after EndoBarrier implantation in comparison with baseline. Medications were classified as "decreased" if the dose of one or more oral agents was lowered or one or more agents were discontinued at the time of treatment completion in comparison with baseline. For subjects in which the dose of one oral glucose-lowering agent was increased and another agent decreased, the change in medications was classified as "not assessable."
Time Frame: Baseline to 52 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Increase in Glucose-Lowering Meds at Week 52: Subjecst who completed 12 month implant duration
- Decrease in Glucose-Lowering Meds; No Change in Glucose-Lowering Meds at Week 52: Subjects who completed 12-month implant duration
Arm/Group | Increase in Glucose-Lowering Meds at Week 52 | Decrease in Glucose-Lowering Meds | No Change in Glucose-Lowering Meds at Week 52
Number analyzed (Participants) | 16 | 16 | 16
Participants | 9 | 0 | 7

3. Secondary Outcome: Total Weight Change (kg) at Week 52 Compared to Baseline Weight
Time Frame: Baseline to 52 weeks
Measure: Mean (Standard Deviation); unit: kg
Groups:
- EndoBarrier Liner Device: 52 week treatment of EndoBarrier Liner
Arm/Group | EndoBarrier Liner Device
Number analyzed (Participants) | 16
kg | -6.3 (4.05)

4. Other Pre Specified Outcome: Fasting Plasma Glucose Over Time for All Subjects
Time Frame: Baseline to 12 months post Device Explant
Population: Subjects with a Successful Device Implant Procedure
Measure: Median (Full Range); unit: mmol/L
Arm/Group | Diabetes
Number analyzed (Participants) | 20
mmol/L
  Baseline | 10.9 [5.8 to 16.6]
  Month 3: number analyzed (Participants) | 19
  Month 3 | 7.3 [3.7 to 13.2]
  Month 6: number analyzed (Participants) | 19
  Month 6 | 7.5 [5.4 to 11.9]
  Month 9: number analyzed (Participants) | 17
  Month 9 | 7.6 [5.5 to 11.4]
  Month 12: number analyzed (Participants) | 16
  Month 12 | 7.6 [4.9 to 14.0]
  3 Months Post-Explant: number analyzed (Participants) | 17
  3 Months Post-Explant | 7.4 [3.3 to 10.9]
  6 Months Post-Explant: number analyzed (Participants) | 17
  6 Months Post-Explant | 8.3 [5.2 to 13.6]
  12 Months Post-Explant: number analyzed (Participants) | 17
  12 Months Post-Explant | 8.9 [5.8 to 16.6]

ADVERSE EVENTS:
Groups:
- EndoBarrier Liner Device: All subjects who had a device attempted to be implanted. N = 23
Arm/Group | EndoBarrier Liner Device
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 22/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoBarrier Liner Device (N=23)
Abdominal pain (Gastrointestinal disorders) | 13 (26)
Abdominal pain upper (Gastrointestinal disorders) | 13 (36)
Abdominal pain lower (Gastrointestinal disorders) | 9 (17)
Abdominal distension (Gastrointestinal disorders) | 8 (10)
Diarrhea (Gastrointestinal disorders) | 8 (14)
Nausea (Gastrointestinal disorders) | 8 (10)
Vomiting (Gastrointestinal disorders) | 7 (8)
Flatulence (Gastrointestinal disorders) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 5 (5)
Asthenia (General disorders) | 3 (3)
Hypersensitivity (Immune system disorders) | 2 (2)
Procedural vomiting (Injury, poisoning and procedural complications) | 3 (3)
Nasopharyngitis (Infections and infestations) | 5 (6)
Influenza (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Procedural nausea (Injury, poisoning and procedural complications) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 17 (173)
Iron deficiency (Metabolism and nutrition disorders) | 15 (29)
Headache (Nervous system disorders) | 5 (6)
Somnolence (Nervous system disorders) | 2 (2)
Depression (Psychiatric disorders) | 3 (5)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Hypertension (Vascular disorders) | 2 (4)
Ischemic limb pain (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No